CLINICAL TRIAL: NCT06726811
Title: Low-Dose Droperidol and Its Association with QTc Interval Changes in Emergency Department Patients
Brief Title: Droperidol and QTc Interval Changes in ED Patients
Status: Recruiting | Type: Observational
Sponsor: CHRISTUS Health (Other)
Responsible Party: Principal Investigator, Aaron Bartoe, Principal Investigator, CHRISTUS Health
Other Study IDs: 2025-026
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Emergency Department Patient; QTc Intervals Changes
Keywords: Droperidol; QTc Interval Changes; Emergency Department Patients
MeSH Terms: interventions — Droperidol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Droperidol injection — 2.5 mg

SUMMARY:
Objectives To assess the association of low-dose Droperidol administration in the emergency department with changes in the QTc interval.

Hypothesis Our study is designed to test the null hypothesis that there will be no clinically significant change in QTc interval after administration of 2.5mg of IV Droperidol during an emergency department visit.

DETAILED DESCRIPTION:
The investigators plan to conduct ECG evaluation for QT interval both before and after patients are given 2.5 mg of droperidol. Specifically, a convenience sample of consenting adult patients, ages 18 years and older, who present to the ED, and are in a cardiac-monitored bed in the ED who, at the discretion of their treating physician, have an ECG recorded and then receive a dose of 2.5 mg of droperidol IV will be enrolled in our study. The investigators will then have a second ECG printed at least 5 minutes and no more than 30 minutes after the droperidol is given. Change in QT interval between the two ECGs will be documented. It may be necessary to review the EMR in order to document the time of droperidol administration.

These post-droperidol ECGs will not be stored in the electronic medical record nor read by a physician in real time. Treatment decisions regarding the patient's medical care in the ED will not be affected by these second ECGs; decisions about whether other ECGs may be needed will be made by the treating physician. The primary study outcome will be the percentage of the study population who experience a clinically significant increase in QTc after low-dose droperidol administration, defined as an increase in QTc of 20 ms or greater. Secondary outcome measures will be the mean change in QTc across the study population, and the percentage of the study population for whom the administration of low-dose droperidol is associated with an increase in QTc that re-classifies them as having a prolonged QTc (>450 ms in men and >470 ms in women).

ELIGIBILITY:
Inclusion Criteria:

* ED patients ages 18 years or older in a cardiovascular-monitored bed who have both an ECG and a 2.5 mg dose of IV droperidol ordered by their treating physician will be eligible for inclusion.

Exclusion Criteria:

* Refusal to provide consent.
* Administration of droperidol before the first ECG is performed.
* Inability to complete the consent form and questionnaire due to clinical instability, severe pain, or disorientation as determined by a study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * The population being studied will be a convenience sample of adult emergency department patients.
  * Eligibility in the study will be based on the treating physician's decision to have administered droperidol and to obtain an ECG - participation in the study will not affect the patient's care.
  * The minimum number of study subjects will be 100.
  * The maximum number of study subjects will be 500.
  * There will be no use of special subject populations.
  * Investigators will also track how many eligible patients refuse to participate. (See "Participation Status" on the survey instrument, Data Collection Form)
  * Written consent will be required for each participant at the top of the survey. (See "Survey Instrument", Data Collection Form)
  * Patients will be enrolled only once.
  * Participants will not receive any form of compensation and will not be billed for the additional ECG.
  * Vulnerable adult populations may be included who are able to give consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
ECG Evaluation | 30 minutes after Droperidol is given.
  We plan to conduct ECG evaluation for QT interval both before and after patients are given 2.5 mg of droperidol.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRISTUS Spohn Hospital Corpus Christi-Shoreline, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] White PF. Droperidol: a cost-effective antiemetic for over thirty years. Anesth Analg. 2002 Oct;95(4):789-90. doi: 10.1097/00000539-200210000-00001. No abstract available. PMID 12351246
- [Background] Trinkley KE, Page RL 2nd, Lien H, Yamanouye K, Tisdale JE. QT interval prolongation and the risk of torsades de pointes: essentials for clinicians. Curr Med Res Opin. 2013 Dec;29(12):1719-26. doi: 10.1185/03007995.2013.840568. Epub 2013 Sep 23. PMID 24020938
- [Background] Pickham D, Helfenbein E, Shinn JA, Chan G, Funk M, Weinacker A, Liu JN, Drew BJ. High prevalence of corrected QT interval prolongation in acutely ill patients is associated with mortality: results of the QT in Practice (QTIP) Study. Crit Care Med. 2012 Feb;40(2):394-9. doi: 10.1097/CCM.0b013e318232db4a. PMID 22001585
- [Background] Nachimuthu S, Assar MD, Schussler JM. Drug-induced QT interval prolongation: mechanisms and clinical management. Ther Adv Drug Saf. 2012 Oct;3(5):241-53. doi: 10.1177/2042098612454283. PMID 25083239
- [Background] Jackson CW, Sheehan AH, Reddan JG. Evidence-based review of the black-box warning for droperidol. Am J Health Syst Pharm. 2007 Jun 1;64(11):1174-86. doi: 10.2146/ajhp060505. PMID 17519460
- [Background] Haddad PM, Anderson IM. Antipsychotic-related QTc prolongation, torsade de pointes and sudden death. Drugs. 2002;62(11):1649-71. doi: 10.2165/00003495-200262110-00006. PMID 12109926
- [Background] Domino KB, Anderson EA, Polissar NL, Posner KL. Comparative efficacy and safety of ondansetron, droperidol, and metoclopramide for preventing postoperative nausea and vomiting: a meta-analysis. Anesth Analg. 1999 Jun;88(6):1370-9. doi: 10.1097/00000539-199906000-00032. PMID 10357347
- [Background] Charbit B, Albaladejo P, Funck-Brentano C, Legrand M, Samain E, Marty J. Prolongation of QTc interval after postoperative nausea and vomiting treatment by droperidol or ondansetron. Anesthesiology. 2005 Jun;102(6):1094-100. doi: 10.1097/00000542-200506000-00006. PMID 15915019
- [Background] Charbit B, Alvarez JC, Dasque E, Abe E, Demolis JL, Funck-Brentano C. Droperidol and ondansetron-induced QT interval prolongation: a clinical drug interaction study. Anesthesiology. 2008 Aug;109(2):206-12. doi: 10.1097/ALN.0b013e31817fd8c8. PMID 18648229
- [Background] Abriel H, Schlapfer J, Keller DI, Gavillet B, Buclin T, Biollaz J, Stoller R, Kappenberger L. Molecular and clinical determinants of drug-induced long QT syndrome: an iatrogenic channelopathy. Swiss Med Wkly. 2004 Nov 27;134(47-48):685-94. doi: 10.4414/smw.2004.10532. PMID 15616901
- [Background] Cole JB, Lee SC, Martel ML, Smith SW, Biros MH, Miner JR. The Incidence of QT Prolongation and Torsades des Pointes in Patients Receiving Droperidol in an Urban Emergency Department. West J Emerg Med. 2020 Jul 2;21(4):728-736. doi: 10.5811/westjem.2020.4.47036. PMID 32726229
- [Background] Fortney JT, Gan TJ, Graczyk S, Wetchler B, Melson T, Khalil S, McKenzie R, Parrillo S, Glass PS, Moote C, Wermeling D, Parasuraman TV, Duncan B, Creed MR. A comparison of the efficacy, safety, and patient satisfaction of ondansetron versus droperidol as antiemetics for elective outpatient surgical procedures. S3A-409 and S3A-410 Study Groups. Anesth Analg. 1998 Apr;86(4):731-8. doi: 10.1097/00000539-199804000-00011. PMID 9539593
- [Background] Hernandez-Rodriguez L, Bellolio F, Cabrera D, Mattson AE, VanMeter D, Grush AE, Oliveira J E Silva L. Prospective real-time evaluation of the QTc interval variation after low-dose droperidol among emergency department patients. Am J Emerg Med. 2022 Feb;52:212-219. doi: 10.1016/j.ajem.2021.12.039. Epub 2021 Dec 22. PMID 34959024
- [Background] Tracz K, Owczuk R. Small doses of droperidol do not present relevant torsadogenic actions: a double-blind, ondansetron-controlled study. Br J Clin Pharmacol. 2015 Apr;79(4):669-76. doi: 10.1111/bcp.12527. PMID 25293524
- [Background] Weibel S, Rucker G, Eberhart LH, Pace NL, Hartl HM, Jordan OL, Mayer D, Riemer M, Schaefer MS, Raj D, Backhaus I, Helf A, Schlesinger T, Kienbaum P, Kranke P. Drugs for preventing postoperative nausea and vomiting in adults after general anaesthesia: a network meta-analysis. Cochrane Database Syst Rev. 2020 Oct 19;10(10):CD012859. doi: 10.1002/14651858.CD012859.pub2. PMID 33075160